CLINICAL TRIAL: NCT06370494
Title: Testing New Models of Diabetes Self-Management to Improve Population Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Marcia G Ory, Regents and Distinguished Professor, Texas A&M University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2020-0956D
Record Dates: First submitted 2024-03-08; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) was conducted to assess the outcomes associated with different technological intervention approaches. This 3-arm RCT assessed independent and combined interventions:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Making Moves with Diabetes [MMWD] Group (Experimental): Virtual asynchronous training and periodic one-on-one counseling with a clinical diabetes educator, either a Registered Nurse (RN) or Registered Dietitian Nutritionist (RDN). The program was recognized by the American Diabetes Association during this study. The intervention included 8 hours of online diabetes education, 30 minute 1:1 virtual education and counseling with a diabetes educator, and 3 and 6-month follow-ups.
  Interventions: Behavioral: Living Healthier with Diabetes
- App Group (Experimental): Smartphone application for more continuous but less structured chat support. This app was recognized by the American Diabetes Association. The intervention included access to online diabetes support tools and ability to message a diabetes specialist for support, and 3 and 6-month follow-ups.
  Interventions: Behavioral: Living Healthier with Diabetes
- Combo Group (Experimental): A combined approach for maximal support and reinforcement. The intervention included 8 hours of online diabetes education, 30 minute 1:1 virtual education and counseling with a diabetes educator, access to the app with online diabetes support tools and ability to message a diabetes specialist for support, and 3 and 6-month follow-ups.
  Interventions: Behavioral: Living Healthier with Diabetes

INTERVENTIONS:
Behavioral: Living Healthier with Diabetes — Interventions are different aspects of digital health utilizing American Diabetes Association recognized diabetes programs/applications or a combined approach. All participants were randomly assigned to their education arm and received an A1c kit, glucometer, testing strips, and surveys.

SUMMARY:
Aim 1.1 To understand if diabetes self-management education and support (DSMES) improves diabetes-related outcomes among those with Type 2 diabetes living in Texas.

Aim 1.2 To examine how rurality affects study participation, engagement in, and effectiveness of different education interventions.

These aims are based on a randomized controlled trial of different evidence-based diabetes self-management interventions.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) was conducted to assess the outcomes associated with different technological intervention approaches. This 3-arm RCT assessed independent and combined interventions:

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM) - self-reported diagnosis by a health care provider
* HbA1c value greater than or equal to 7.5%
* Adults ages 25 years and older
* All genders
* Have access to device (smartphone/tablet which meets iOS 13 or above or similar system requirements/iPhone 7 and above or Android 6 and above) and internet in order to view online diabetes education content
* Ability to read and speak English
* Resides in Texas

Exclusion Criteria:

* Pregnant women
* Participation in ADA-recognized or AADE-accredited diabetes self-management education program lasting at least eight hours within previous six months
* Engagement with ADA-recognized or AADE-accredited smartphone application with certified diabetes educators providing tracking and health coaching within the previous six months
* Those diagnosed with any conditions listed below (determined by self-report): Liver failure, End-stage renal disease (stage 4 or 5), Congestive heart failure (grade C or D), Organ transplant or bone marrow transplant, Cystic fibrosis, Malignant neoplasm or bone marrow transplant
* Criteria excludes individuals based on language. Participants must be able to read and speak English. Technology-based education and support (TBES) is available only in English.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
A1C -Change in HbA1c between baseline, 3 months, and 6 months is the primary outcome. | 12 months
  A1C values will be treated continuously in analyses, with possible values ranging from 4 to 14 due to instrument precision at the higher values.

SECONDARY OUTCOMES:
Diabetes Knowledge: Knowledge of diabetes will be measured by the simplified version of the Revised Diabetes Knowledge Scale (True/False version). | 12 months
  Knowledge of diabetes will be measured by the simplified version of the Revised Diabetes Knowledge Scale (True/False version). 10 True False questions will be included with answers of True, False, and I don't know. Correct responses receive 1 point indicating a range of 0-10 points for this outcome measure.
Diabetes Self Care | 12 months
  Diabetes self-management behavior will be measured by the adapted Summary of Diabetes Self-Care Activities Measure (SDSCA). The SDSCA is a brief self-report questionnaire that includes items assessing the following aspects of the diabetes regimen: general diet, specific exercise, blood-glucose testing, foot care, alcohol, and smoking. The scale has been adapted to examine self-care activities before and since COVID-19. Furthermore, a question about alcohol drinking has been added. Diabetes Self-care is the number of days a participant performed certain activities pertaining to diabetes care in a typical week. The diabetes self care scale is 8 questions asking how many days per week a participant engaged in a behavior on a scale of 0-7 days. Therefore, the scale ranged from 0-56 points, with higher points indicating greater occurrence of diabetes self care.
Diabetes Care Confidence | 12 months
  Confidence in doing specific activities related to diabetes will be measured by the Self-Efficacy for Diabetes Scale. The scale is a self-report instrument that asks how confident individuals feel doing specific activities related to diabetes (e.g., diet, exercise, blood sugar monitoring).Diabetes confidence is how confident a participant is in their own ability to perform certain activities. To analyze this, a sum of 8 questions was taken. Diabetes confidence scale is 8 questions on scale of 1-10 ranging from ("not at all confident" to "totally confident"). The higher the sum is, the higher the confidence. Therefore, final outcome scores will range from 8-80, with higher scores indicating greater confidence in diabetes management.
Diabetes care distress | 12 months
  Distress related to living with diabetes will be measured by the 2-item Diabetes Distress Screening Scale (DDS2). The DDS2 asks participants to rate the degree to which of perceived magnitudes of problems concerning diabetes that may have distressed or bothered participants. Diabetes distress is how distress a participant is in performing activities pertaining to diabetes care. Diabetes distress scale is 6 questions on a scale of 1-6 ranging from ("not a problem" to "a very serious problem"). To analyze this, a sum of 6 questions was taken. The higher the sum is, the more distressed the participant is. Therefore, the scale ranged from 6-36 points, with higher points more diabetes distress.
A1C | 12 months
  -Number of participants with A1c reduction that is at least .5 (clinically significant). In addition to the continuous A1C measurements, an indicator variable will be created to indicate a clinically meaningful change (e.g., whether A1C dropped more than 0.5 at the 6-month). Possible A1c values ranging from 4 to 14 due to instrument precision at the higher values.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Ory, Principal Investigator — Texas A&M Health
Locations (1):
- Texas A&M Health, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No